CLINICAL TRIAL: NCT00377039
Title: A Multi-Centre, Randomised, Double-Blind, Placebo Controlled, Parallel Group Exploratory Study to Investigate the Efficacy, Safety and Tolerability of AD 337 in the Treatment of Fibromyalgia in Female Subjects.
Brief Title: A Multicentre Trial to Determine the Efficacy and Safety of AD-337 in the Treatment of Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sosei (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD337-021
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2007-10-02 (Estimated); Status verified 2007-09

CONDITIONS: Fibromyalgia
Keywords: ACR 1990 Fibromyalgia; Fibromyalgia Impact Questionnaire
MeSH Terms: conditions — Fibromyalgia

INTERVENTIONS:
Drug: AD 337

SUMMARY:
This is a multicentre, randomized, double-blind, placebo controlled, parallel group exploratory study to investigate the efficacy, safety and tolerability of AD 337 in the treatment of fibromyalgia in female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-65
* Meet ACR 1990 criteria for classification of Fibromyalgia
* Able and willing to discontinue CNS active therapies

Exclusion Criteria:

* If pain is NOT primarily due to Fibromyalgia
* Current or prior history of serious psychiatric disorder
* Pregnant/breastfeeding
* QTc > 470ms
* Failure to respond to 2 or more adequate regimes of different classes of antidepressants.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-08; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
The Fibromyalgia Impact Questionnaire total score after 4 weeks treatment

SECONDARY OUTCOMES:
These will be
FIQ Total score at weeks 1, 2, 3, at end of study and overall
FIQ subscales at weeks 1, 2, 3, 4 at end of study and overall
Short form McGill Pain questionnaire subscales at weeks 1, 2, 3, 4 at end of study and overall
Tender point assessment (ACR 1990 criteria) scores at weeks 2, 4 at end of study and overall
Hospital Anxiety and Depression Scale subscales at weeks 2, 4 and overall
Fibromyalgia Health Assessment Questionnaire total score at weeks 1, 2, 3, 4 at end of study and overall

CONTACTS AND LOCATIONS:
Overall Officials: David L Scott, Principal Investigator — King's College London
Locations (1):
- David L Scott, London, United Kingdom